CLINICAL TRIAL: NCT06763965
Title: A Phase Ib/Ⅱ Clinical Study to Evaluate the Safety, Tolerability, Biodistribution Characteristics and Preliminary Efficacy of Recombinant Human nsIL12 Oncolytic Adenovirus Injection (BioTTT001) in Patients With Recurrent/Progressive High-grade Glioma.
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of BioTTT001 in Patients With Recurrent/Progressive High-grade Glioma.
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Bio-Targeting Therapeutics Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJCT-01-102
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Recurrent High-grade Glioma
Keywords: Oncolytic virus; IL-12; Adenovirus
MeSH Terms: conditions — Glioma; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioTTT001 injection (Experimental): BioTTT001 is administered as a multiple Intratumoral injection. The dose groups to be infusion were 1.0×10^10 viral particle (VP) ,5.0×10^10 VP and 2.5×10^11 VP based on the 3+3 dose escalation principle.
  Interventions: Biological: BioTTT001 injection

INTERVENTIONS:
Biological: BioTTT001 injection — BioTTT001 is administered as a multiple Intratumoral injection. The dose groups to be infusion were 1.0×10^10 viral particle (VP) ,5.0×10^10 VP and 2.5×10^11 VP based on the 3+3 dose escalation principle.

SUMMARY:
This study is a single-arm, open-label, dose-escalation and dose-expanding Phase Ⅰb/Ⅱ clinical study to evaluate the safety, tolerability, biodistribution characteristics and preliminary efficacy of recombinant human nsIL12 oncolytic adenovirus injection (BioTTT001) in patients with recurrent/progressive high-grade glioma.

DETAILED DESCRIPTION:
Phase Ⅰb Dose Escalation Study:Three dose groups were established in the dose escalation phase, namely 1.0×10^10 VP, 5.0×10^10 VP and 2.5×10^11 VP. The traditional "3+3" dose escalation method was used for dose escalation, with at least 3 subjects enrolled in each dose group, and each subject received only one corresponding dose until the MTD and/or RP2D were determined.It is planned to enroll 12~18 subjects, and the final sample size of enrollment depends on the number of DLT, the number of dose groups that are escalated before the DLT is observed, and the determination of the MTD.

Phase Ⅱ Dose Expansion Study:In this phase, one dose group was selected for a dose expansion study to further evaluate the efficacy and safety of BioTTT001 in patients with recurrent/progressive high-grade glioma.It is planned to select 1 dosage that may be used for phase Ⅰ clinical research to expand enrollment, and it is planned to enroll 10~30 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old (including the critical value), male or female;
2. Patients with high-grade glioma who have recurred/progressed after receiving standard therapy as confirmed by histopathological confirmation meeting the 2021 World Health Organization (WHO) classification criteria for central nervous system tumors;
3. Karnofsky Performance Score (KPS) ≥ 60 points (see Appendix 2);
4. Suitable for placement of Ommaya sac as judged by the investigator to be eligible for administration;
5. Estimated survival ≥ 3 months;
6. Good organ function;
7. Voluntary participation and ability to sign informed consent form prior to the start of study-related procedures, after explaining the content of the study;
8. Subjects of childbearing potential and sexually active partners must be willing to use a medically approved and effective method of contraception, such as a double-barrier method of contraception, during treatment and for 6 months after the last dose, and the male agrees not to donate sperm;
9. Females of childbearing potential, must have a negative blood pregnancy test result within 7 days prior to the first dose and be willing to undergo additional pregnancy tests during the study. Females of childbearing potential who have not undergone surgical sterilization (i.e., bilateral tubal ligation, bilateral oophorectomy, or total hysterectomy) or are not postmenopausal; Menopause is the absence of menopause for 12 months in women over ≥ age of 45 and the exclusion of other causes of amenorrhea. In addition, serum follicle-stimulating hormone (FSH) levels in women under 50 years of age must be in the postmenopausal range for menopause to be confirmed;
10. Good compliance, willing and able to follow all research procedures, and cooperate with observation and follow-up.

Exclusion Criteria:

1. Received anti-tumor drug therapy such as radiotherapy, chemotherapy, biological therapy, endocrine therapy, targeted therapy and other anti-tumor drugs within 4 weeks before the first dose (excluding immunotherapy, nitrosourea, mitomycin C, oral fluorouracil, small molecule targeted drugs, and traditional Chinese medicines with anti-tumor indications);
2. Treatment with any other unmarketed investigational drug within 4 weeks prior to the first dose;
3. Surgical surgery of major organs within 4 weeks prior to the first dose (excluding live puncture) or have had significant trauma, or need to undergo elective surgery during the study;
4. Those who have a history of cell therapy, gene therapy, and oncolytic virus therapy in the past;
5. Those who have known or suspected hypersensitivity to the active ingredients of the study drug, excipients, and imaging contrast agents;
6. Those who have a history of organ transplantation or plan to undergo organ transplantation during the study;
7. Patients with active infection or uncontrollable infection requiring intravenous systemic therapy, or fever of unknown cause > 38.5°C during the screening period and before the first dose;
8. Accompanied by severe coagulation disorder or other evidence of obvious bleeding risk; history of gastrointestinal bleeding; Any other ≥ CTCAE grade 2 bleeding event within the past 6 months;
9. Patients with herniation syndrome;
10. Pregnant or lactating females.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 28 days within BioTTT001 injection
  The incidence and severity of all types of adverse events evaluated based on NCI-CTCAE5.0
DLT、MTD and/or RP2D | 28 days within BioTTT001 injection
  Maximum tolerated dose (MTD)、Dose-limiting toxicity（DLT）、Recommended Phase II Dose（RP2D）
OS12 | 12 months
  12-month survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Sanbo Brain Hospital, Capital Medical University, Beijing, Haidian District, China